CLINICAL TRIAL: NCT07354945
Title: An Evaluation of Visual Comfort, Adaptation and Overall Satisfaction in Myopic Children Using A.M.L. Series of Lenses
Brief Title: An Evaluation of Myopia Control Lenses on Wearing Experience in Myopic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WS10450
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A.M.L. Series of Lenses (Experimental)
  Interventions: Device: A.M.L. Series of Lenses

INTERVENTIONS:
Device: A.M.L. Series of Lenses — Participants will be wearing A.M.L. series of lenses for a period of 2 weeks.

SUMMARY:
The goal of this research study is to understand the wearing experience of A.M.L. series of lenses in myopic children. The main questions it aims to answer are:

* How quickly and effectively children adapt to the A.M.L. series of lenses?
* The proportion of children who adapted to the A.M.L. series of lenses within 4 to 6 days?

  40 myopic children aged 6 to 12 years will be recruited as participants, and all of them will be wearing A.M.L. series of lenses.

Participants will:

* Wear A.M.L. series of lenses for a period of 2 weeks
* Visit at day 4-6, week 1 and week 2.

DETAILED DESCRIPTION:
Myopia prevalence among Chinese children has increased markedly in recent years, representing a major public health concern. As myopia management options expand, expectations have shifted beyond efficacy alone to include wearing comfort, adaptation, and visual quality. Spectacle lenses remain the primary modality for myopia correction and play a critical role in daily visual experience. Optical defocus-based spectacle lenses with microlens designs have demonstrated efficacy in slowing myopia progression. Although existing studies have reported on the adaptation of spectacle lenses incorporating microlens designs, there are currently no data available for the A.M.L. series of lenses. This study aims to evaluate adaptation, wearing comfort, and user satisfaction with the A.M.L. series spectacle lenses.

This is a one arm, prospective, interventional study, it will include 40 children, with adaptation, comfort, and satisfaction evaluated after 4 days, 1 week, and 2 weeks of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer participant
* Informed consent of parent/guardian and assent of participant
* Age equal to or greater than 6 years and not older than 12 years at the time of signing informed consent and assent
* Spherical equivalent refraction (SER) by cycloplegic autorefraction equal or less than -0.50 D and equal or greater than -4.75D with astigmatism not more than 2.00 D on both eye
* Difference in SER (anisometropia) between two eyes should not exceed 1.50 D
* Best corrected visual acuity (BCVA) better than or equal to +0.10 LogMAR in each eye
* Be in good general health, based on the participant and the parent's/guardian's knowledge
* Willingness and ability to participate in study and comply with all scheduled visits

Exclusion Criteria:

* History of Atropine, Orthokeratology, or Red Light treatment
* Strabismus by cover test at near or distance wearing correction
* Amblyopia
* Any ocular or systemic condition known to affect refractive status (e.g. keratoconus, diabetes, Downs syndrome, or other developmental disorders, etc.)
* Current use of ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state
* History of ocular injury or surgery
* Participation in any clinical study within 30 days of the Baseline visit
* Study participants deemed inappropriate for the study by the investigator
* The inherent ocular/systemic discomfort (dry eyes, visual fatigue, headaches, etc.) that may affect the evaluation of the study lens wearing experience, from the investigator's perspective

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
The proportion of children who adapted to the study lenses within 4 to 6 days without reporting any symptoms. | Day 6

SECONDARY OUTCOMES:
Proportions of children who adapted within 1 day | Day 4-6
Mean wearing time per week and per day | Week 2
Activity-specific visual comfort using questionnaire at 4-day and 2-weeks | Day 4-6, Week 2
  Visual Comfort in Different Activities Questionnaire (5-point Likert scale, range 1-5). For negatively worded items, higher score indicate worse visual comfort, whereas positively worded items, higher score indicate better visual comfort.
Overall satisfaction reported at 4 days and 2 weeks | Day 4-6, Week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Meishimeijing Ophthalmology Clinic Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drobe B, Yang A, Huang Y, et al. Adaptation and visual comfort in children with new spectacle lenses containing concentric rings of contiguous aspherical micro-lenses for myopia control. Investigative Ophthalmology & Visual Science June 2020, Vol.61, 94.